CLINICAL TRIAL: NCT05367648
Title: The Effect of Protein Hydrolysate Supplementation to Influence the Expression of Systemic Muscle Function Markers Following Resistance Type Exercise in Male Subjects
Brief Title: Effects of Protein Hydrolysate Supplement on Systemic Muscle Function Markers Following Resistance Type Exercise in Male Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nuritas Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PN20.004-INTERNAL
Record Dates: First submitted 2022-03-25; First posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Muscle Injury
Keywords: muscle; function; markers; resistance; exercise; protein; hydrolysate; supplement; Elio
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elio (supplement under investigation) (Experimental): 3g of Elio administered orally daily with the first meal of the day for a 17 day period
  Interventions: Dietary Supplement: Elio
- Place (Placebo Comparator): 3g of SMCC administered orally daily with the first meal of the day for a 17 day period
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Elio — Elio™ supplementation, a protein hydrolysate derived from fava bean protein extract
  Arms: Elio (supplement under investigation)
Other: Placebo — Placebo comparator
  Arms: Place

SUMMARY:
The effect of exercise on serum concentrations of creatine kinase (CK) and subsequent use of protein hydrolysate supplementation, Elio, to influence the expression of CK following resistance type exercise in male subjects. A two subject trial of Elio administered 3 grams per day in assessing its effects on post-exercise increases in markers associated with muscle injury and exertion

DETAILED DESCRIPTION:
Following muscle injury or exertion, several muscle specific enzymes (CK, LDH), metabolites (Acylcarnitine, FFAs) and inflammatory cytokines (IL-6, CRP) display a temporal increase in expression over 24-96hrs. For example, the muscle specific isoform of CK has been demonstrated to be elevated in the serum of subjects following eccentric resistance training with increased expression from 3hrs post exercise with a peak between 72 hrs and 96 hrs post exercise and up to 120 hrs post exercise.

Similarly, post training muscle homeostasis and injury is also associated with the infiltration of white blood cell populations namely macrophages and neutrophils, this increase in infiltration is accompanied by increases in the expression of inflammatory cytokines such as IL-6 and Il-8.

Specifically, the interleukin IL-6, has been found to be increased in concentration by up to 10-fold, compared to pre-exercise baseline, when subjects complete knee extension, cardio-vascular or eccentric exercise-based routines. Similar post-exercise or injury related increases in markers such as CRP and LDH have also been identified.

While these processes form part of the natural biological processes underpinning muscle and homeostasis, excessive or chronic elevation of these factors can prolong recovery, exacerbate injury and impair performance. Therefore, developing natural interventions that enhance or augment muscle homeostasis, reduce the likelihood of muscle injury and suppress excessive post-exercise inflammatory responses (IL-6, CRP), to enhance recovery would be highly desirable.

Several studies have been conducted where the effect of naturally derived compounds or milk-based products have been explored. Recent analysis of bovine colostrum in lower-division football players demonstrated that 3g supplementation over a 6-week period could significantly reduce the expression of markers such as CK, CRP and IL-6 following Loughborough Intermittent Shuttle Tests.

This reduction in systemic markers induced by the supplementation also corresponded to an improved performance in this routine as compared to subjects receiving 3g of whey supplementation. Resistance type exercise represents an effective model to examine the effects of injury on this panel of markers and is a controlled experimental condition to investigate the efficacy of supplementation on both performance and underlying biochemical processes.

Nutritional strategies to improve post-exercise blood marker profiles are scarce, but there is evidence that the right strategy can be effective both in females and males across a lifespan.

Resistance exercise (1-RM) routines in elderly female subjects have been shown to induce increases in IL-6 and CRP; studies also show that whey supplementation can assist in suppressing post-exercise increases in IL-6. Furthermore, male endurance athletes (aged 18-45 yrs) that supplemented with DHA and EPA showed significant decreases in circulating IL-6 and CK concentrations post-isokinetic testing compared to pre-supplementation.

Therefore, it is important for this study to examine the effects of Nuritas' Elio™ product on post-resistance exercise increases in these key markers of muscle fatigue and injury.

Given the essential role of NAD+ in the regulation of multiple cellular processes known to contribute to age-related decline in cellular function (metabolic homeostasis, DNA damage repair and sirtuin activity), investigators sought to ascertain whether increased pAMPK seen upon in vitro Elio administration translated into an increase in intracellular NAD+ concentration as measured by HPLC.

Preliminary data suggested that treatment of primary human fibroblasts with Elio resulted in a statistically significant increase (p<0.05) in intracellular levels of NAD+ relative to control (mean increase of 17%, ± 6.421 S.E.M., n=4). Given the significant increase in intracellular NAD+ concentration observed in vitro following short-term Elio treatment, longer-term Elio administration in vivo was assessed as a secondary endpoint.

7.2 Introduction

The benefits of regular and routine physical activity and exercise are well documented. Frequent physical activity are necessary tools in preventing modern life-style associated diseases such as type II diabetes, obesity and other cardio-vascular conditions. Nonetheless, injuries resulting from physical activity can have a profound impact on individuals' quality of life and work-place productivity. Periods of intense physical activity and exertion can lead to disruption of normal muscle homeostasis. Resultant muscle injury and recovery can impact upon quality of life especially in adult populations. Socio-economic studies have indicated that common skeletal-muscular injuries commonly encountered by male and female populations during regular exercise account for nearly 49% of work-place absences and 60% of permanent work incapacity. Taking this into account, studies have estimated the cost of these injuries to be in excess of €200bn due to enforced absence and lack of productivity.

It is therefore important to develop products that can lessen the impact of these injuries, which individuals succumb to or expedite their recovery

ELIGIBILITY:
Inclusion Criteria:

* Participants agree to comply with study procedures
* Participants agree to abstain from taking additional supplements throughout the testing period, with particular emphasis placed upon protein-based products
* Participants agree to maintain their normal diet and exercise routine throughout the study
* BMI between 18.5 to 29.9 kg/m2
* Participants agree to refrain from consuming alcohol in the 48 hrs leading up to a test day
* Willingness to complete questionnaires, records and diaries associated with the study and to complete all clinic visits
* Provide voluntary, written, informed consent to participate in the study.
* Refrain from any sort of exhaustive physical exercise from 48 hrs prior to each test.
* Healthy as determined by medical examination at screening visit
* Willingness to complete food diaries (including two weekdays and one weekend day the week before testing) dietary intake records shall be completed before and during the study
* Non-smoker
* Subjects must possess a smart phone

Exclusion Criteria:

* .Alcohol or drug abuse in past year
* Participation in any other clinical trial in the last 3 months from time of randomisation
* Subject has a known allergy to the test material's active or inactive ingredients
* Subjects with unstable medical conditions
* Clinically significant abnormal laboratory results at screening
* Any complaints that could interfere with ability to exercise
* Individuals who are cognitively impaired and/or who are unable to give informed consent
* Any co-morbidities interacting with mobility or muscle metabolism of the lower limbs (e.g., arthritis, spasticity/rigidity, all neurological disorders and paralysis)
* Creatine supplements, anticoagulants, corticosteroids, growth hormones, testosterone, immunosuppressants, or exogenous insulin over the previous six months
* Presence or history of neurological disorders or significant psychiatric illness
* Any other condition which in the Investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject
* Participation in resistance or aerobic exercise within 48 hours of Day 0, Day 4, Day 15 and Day 19 visits in this trial
* Have been in contact with a suspected or confirmed case of Covid-19 in the previous 14 days
* Are Hepatitis A or B positive, HIV positive or have had a sexual partner who is infected with hepatitis or HIV

Ages: 30 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 2 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2020-10-09 (Actual); Study Completion 2020-11-24 (Actual)

PRIMARY OUTCOMES:
Induction of creatine kinase (CK) across a range of time points | 19 days
  Induction of detectable concentrations of CK in response to exercise induced muscle damage

SECONDARY OUTCOMES:
Attenuation of post-resistance exercise increases in serum CK | 19 days
  Attenuation of post-resistance exercise alterations in markers related to muscle homeostasis compared to Baseline at Day 4, Day 15 and Day 19

OTHER OUTCOMES:
Alterations in plasma IL-6 as a marker related to muscle homeostasis/inflammation compared to Baseline | 19 days
  Secondary objective
Change in whole blood NAD+ (as a marker of metabolism) compared to baseline | 19 days
  Secondary objective

CONTACTS AND LOCATIONS:
Overall Officials: Brian Keogh, Principal Investigator — Nuritas Ltd
Locations (1):
- Nuritas Ltd, Dublin, Leinster, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baird MF, Graham SM, Baker JS, Bickerstaff GF. Creatine-kinase- and exercise-related muscle damage implications for muscle performance and recovery. J Nutr Metab. 2012;2012:960363. doi: 10.1155/2012/960363. Epub 2012 Jan 11. PMID 22288008
- [Background] Minetto MA, Rainoldi A, Gazzoni M, Ganzit GP, Saba L, Paccotti P. Interleukin-6 response to isokinetic exercise in elite athletes: relationships to adrenocortical function and to mechanical and myoelectric fatigue. Eur J Appl Physiol. 2006 Nov;98(4):373-82. doi: 10.1007/s00421-006-0285-7. Epub 2006 Sep 2. PMID 16951949
- [Background] Calle MC, Fernandez ML. Effects of resistance training on the inflammatory response. Nutr Res Pract. 2010 Aug;4(4):259-69. doi: 10.4162/nrp.2010.4.4.259. Epub 2010 Aug 31. PMID 20827340
- [Background] Kotsis V, Grassi G. The enigma of obesity-induced hypertension mechanisms in the youth. J Hypertens. 2016 Feb;34(2):191-2. doi: 10.1097/HJH.0000000000000829. No abstract available. PMID 26682787
- [Background] Benito PJ, Cupeiro R, Ramos-Campo DJ, Alcaraz PE, Rubio-Arias JA. A Systematic Review with Meta-Analysis of the Effect of Resistance Training on Whole-Body Muscle Growth in Healthy Adult Males. Int J Environ Res Public Health. 2020 Feb 17;17(4):1285. doi: 10.3390/ijerph17041285. PMID 32079265
- [Background] Nabuco HCG, Tomeleri CM, Fernandes RR, Sugihara Junior P, Cavalcante EF, Cunha PM, Antunes M, Nunes JP, Venturini D, Barbosa DS, Burini RC, Silva AM, Sardinha LB, Cyrino ES. Effect of whey protein supplementation combined with resistance training on body composition, muscular strength, functional capacity, and plasma-metabolism biomarkers in older women with sarcopenic obesity: A randomized, double-blind, placebo-controlled trial. Clin Nutr ESPEN. 2019 Aug;32:88-95. doi: 10.1016/j.clnesp.2019.04.007. Epub 2019 May 13. PMID 31221297
- See also: Muscle and Joint Pain Costs European Economies Billions in Time and Money — https://www.ehstoday.com/health/article/21908653/muscle-and-joint-pain-costs-european-economies-billions-in-time-and-money